CLINICAL TRIAL: NCT01672125
Title: Effect of Upper Limb Posture on Limb Volume as Expressed in Circumference Measurement in Healthy Women and in Women With Breast Cancer Related Lymphedema
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: TASMC-12-EG-449-CTIL
Record Dates: First submitted 2012-08-21; First posted 2012-08-24 (Estimated); Last update posted 2012-08-24 (Estimated); Status verified 2012-08

CONDITIONS: Breast Cancer; Lymphedema
MeSH Terms: conditions — Breast Neoplasms; Lymphedema

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- women who have completed treatments: women who have completed breast cancer treatments, with a diagnosis of unilateral arm lymphedema, in the intensive phase of lymphedema treatment
  Interventions: Other: circumferential measurements in different upper limb positions.
- women who have completed treatment in maintenance phase: women who have completed breast cancer treatment and are in the maintenance phase of lymph edema treatment
  Interventions: Other: circumferential measurements in different upper limb positions.
- healthy women: healthy women adjusted in age and BMI
  Interventions: Other: circumferential measurements in different upper limb positions.

INTERVENTIONS:
Other: circumferential measurements in different upper limb positions. — circumferential measurements in different upper limb positions, in 90 degrees forward flexion and depending position

SUMMARY:
Lymphedema is one side effect of breast cancer treatment. Measuring the edematous limb enables monitoring changes in the lymphedema and the effect of treatment. Circumference measurement using a measuring tape is an inexpensive simple method and therefore useful and widespread in clinical practice. Circumference measurement performance varies amongst therapists and lacks uniformity in the literature. To date, the effect of different limb positions on measurement results has not been examined.

Purpose: The purpose of this study is to describe 1) the effect of position on upper limb volume measurement by using circumference measurement and 2) to examine whether the difference between positions are similar in the upper limbs of the same woman, and 3) between groups of women who are in the intensive phase, in the maintenance phase of lymphedema treatment and women without lymphedema

DETAILED DESCRIPTION:
Study design: Analytical cross section study Population: Inclusion criteria: 15 women who have completed breast cancer treatments, with a diagnosis of unilateral arm lymphedema, in the intensive phase of lymphedema treatment; 15 women who have completed breast cancer treatment and are in the maintenance phase of lymph edema treatment and 15 healthy women adjusted in age and BMI. Exclusion criteria: active cancer, cardiovascular disorder, wounds or inflammation in the measured upper limb, and illness with fever.

Research tools: Questionnaire to gather personal details, information about the cancer and the lymphedema. Plastic, retractable measuring tape with an accuracy of 1 mm. Fixed points on the limb are measured according to anatomical landmarks and afterwards the limb volume is calculated using the formula for a truncated cone.

ELIGIBILITY:
Inclusion Criteria:

* 15 women who have completed breast cancer treatments, with a diagnosis of unilateral arm lymphedema, in the intensive phase of lymphedema treatment;
* 15 women who have completed breast cancer treatment and are in the maintenance phase of lymph edema treatment and
* 15 healthy women adjusted in age and BMI.

Exclusion Criteria:

* active cancer,
* cardiovascular disorder,
* wounds or inflammation in the measured upper limb, and
* illness with fever.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: women who have completed breast cancer treatments, with a diagnosis of unilateral arm lymphedema, in the intensive phase and in the maintenance phase of lymphedema treatment, 15 healthy women adjusted in age and BMI.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2012-11

PRIMARY OUTCOMES:
Circumferential upper limb measurement | 3 hours for each subject

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Medical Center, Tel Aviv, Israel